CLINICAL TRIAL: NCT05266846
Title: Bevacizumab and Chemotherapy With or Without Pembrolizumab in First Line Alectinib Failed ALK-rearranged Advanced Lung Adenocarcinoma Patients With Persistent 5'ALK: A Phase II Randmized Control Trial
Brief Title: Pembrolizumab Plus Bevacizumab and Chemotherapy for ALK-rearranged NSCLC With Persistent 5'ALK
Acronym: BEYOND
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Deputy Director of Thoracic Oncology Department, Hunan Province Tumor Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022017
Record Dates: First submitted 2022-02-18; First posted 2022-03-04 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: ALK Gene Mutation; Lung Adenocarcinoma; Immunotherapy
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — pembrolizumab; Pemetrexed; Bevacizumab; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab plus Bevacizumab and Chemotherapy (Experimental): Pembrolizumab Plus Bevacizumab and Chemotherapy was used for ALK-rearranged NSCLC With Persistent 5'ALK.
  Interventions: Drug: Pembrolizumab injection
- Bevacizumab plus Chemotherapy (Experimental): Bevacizumab plus Chemotherapy was used for ALK-rearranged NSCLC With Persistent 5'ALK.
  Interventions: Drug: Pembrolizumab injection

INTERVENTIONS:
Drug: Pembrolizumab injection — Pembrolizumab 20mg ivgtt once every 21day Platium based Chemotherapy ivgtt once every 21day Bevacizumab 15mg/kg ivgtt once every 21day
  Other Names: pemetrexed; Bevacizumab; CISPLATIN

SUMMARY:
This is an open-label, multiple centers, two-arms phase II study to evaluate the safety and efficacy Pembrolizumab,Bevacizumab in combination with Chemotherapy could improve PFS in Alectinib Failed ALK-rearranged Advanced Lung Adenocarcinoma with Persistent 5'ALK. The eligible patients should have Stage IV Adenocarcinoma ALK-rearranged tested by NGS Perisitent with 5'ALK Failed from first line Alectinib. The patients should meet the physical requirements to receive Pembrolizumab, Bevacizumab with Chemotherapy. All the patients who meet these requirements will be enrolled in this study. The eligible patients will be treated with Pembrolizumab 200 mg intravenously (IV) plus Bevacizumab 15mg/kg+ Pemetrexed 500mg/m2+Carboplatin AUC=4 for up to 4 cycles followed by Pembrolizumab 200mg Q3W+ Bevacizumab 15mg/kg+Pemetrexed 500mg/m2 for up to 31cycles or until disease progression, intolerable toxicity, or physician or participant decision.

DETAILED DESCRIPTION:
This is an open-label, multiple centers, two-arms phase II study to evaluate the safety and efficacy Pembrolizumab,Bevacizumab in combination with Chemotherapy could improve PFS in Alectinib Failed ALK-rearranged Advanced Lung Adenocarcinoma with Persistent 5'ALK. The eligible patients should have Stage IV Adenocarcinoma ALK-rearranged tested by NGS Perisitent with 5'ALK Failed from first line Alectinib. The patients should meet the physical requirements to receive Pembrolizumab, Bevacizumab with Chemotherapy. All the samples were collected for single-RNA sequencing and DSP to evalutate the TME to predict the efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age on day of signing informed consent.

  * Stage IV ALK-rearranged Lung Adenocarcinoma Persistent with 5'ALK Failed from first line Alectinib

    * Have at least 1 lesion that meets the criteria for being measurable, as defined by RECIST 1.1, and is appropriate for selection as a target lesion, as determined by local site investigator radiology review. Lesions that appear measurable, but have undergone palliative irradiation, cannot be target lesions ④20 FFPE sliders prepared,Subjects who do not have histology samples (defined as core or excisional biopsy, or resections) will need to undergo a new biopsy to provide a tissue sample ⑤Eastern Cooperative Oncology Group performance status 0 or 1

      * Life expectancy ≥3 months

        * Adequate hematologic and end organ function

Exclusion Criteria:

Cancer-Specific Exclusions:

①Active or untreated central nervous system metastases

②Malignancies other than NSCLC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome

General Medical Exclusions:

* Pregnant or lactating women.

  * Has active autoimmune disease that has required systemic treatment in the past 2 years.

    * History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.

      * Positive test for human immunodeficiency virus.

        ⑤Active hepatitis B or hepatitis C.

        ⑥Severe infection within 4 weeks prior to randomization .

        ⑦Significant cardiovascular disease.

        ⑧Illness or condition that interferes with the participant's capacity to understand, follow and/or comply with study procedures.

        ⑨Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment for another health-related problem.

Exclusion Criteria Related to Medications: Prior treatment with anti-programmed death-1, anti-PD-L1 therapeutic antibodies，and anti-VEGF agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2026-11-16 (Estimated); Study Completion 2027-02-16 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years
  Defined as the time from the beginning of treatment to the first imaging disease progression or death (whichever occurs first)

SECONDARY OUTCOMES:
ORR | 2 years
  Defined as the proportion of subjects in complete remission (CR) and partial remission (PR) to the total subjects
DCR | 2 years
  Defined as the proportion of subjects with complete remission (CR), partial remission (PR) and stable disease (SD) to the total subjects

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang C Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China